CLINICAL TRIAL: NCT02529436
Title: Overuse of Antidepressant in Patients With Alzheimer Disease and Associated Disorders : An Observational Study
Brief Title: Overuse of Antidepressant in Patients With Alzheimer Disease
Acronym: OVADAD
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AD2015
Record Dates: First submitted 2015-07-28; First posted 2015-08-20 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Alzheimer Disease
Keywords: overuse antidepressant; dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Near 40% of French people aged 65 years and over and suffering from Alzheimer disease and associated disorders (ADAD) are exposed to antidepressants (AD) versus 13% of those without ADAD. If depression and anxiety disorders are comorbidities frequently associated with dementia, such level of AD exposure suggests an overuse of AD in this population.

Hypothesis: Overuse of AD is frequent in patients with ADAD. It is possible to assess overuse associated with off label prescriptions (no validated indication and excess in prescription duration) Main objective: to assess the prevalence of AD overuse associated with off label prescriptions (no validated indication and excess in prescription duration) in patients aged 70 years and over with ADAD.

Secondary objectives:

1. To assess the prevalence of AD prescribed for a non validated indication
2. To assess the prevalence of AD prescribed with excess in prescription duration
3. To assess the prevalence of psychotropic coprescription and notably the prevalence of the neurologic iatrogenic alerts as defined by the French National Authority for Health
4. To assess factors associated to AD overuse Method: A transversal monocentric study in the geriatric day Bretonneau unit will be performed. Study will be proposed to all eligible patients (with non-opposition of the patient or of his legal representative to the collection of his personal data). Included people will have no supplementary clinical or complementary investigations. The geriatrician in charge will have to systematically collect the indication and the history of the AD treatment. At the end of the evaluation performed in the geriatric day unit, the geriatrician will have to conclude to the AD overuse or not associated with off label prescription. Doubtful case will be examined by a validation committee.

Eligibility criteria: Patient consulting in geriatric day hospital with age ≥70 years and dementia according to DSMIV criteria, whatever its level and antidepressant prescription.

Sample size Considering that 40% of people suffering from ADAD are prescribed antidepressant (data from French Health Insurance), the number of eligible patients consulting in the geriatric day swill be 65 in 6 months. If 10% of them are opposed to the collection of their personal data and if the overuse of AD is near 50%, precision of the result will be 12.8% (95%CI bilateral).

Duration of inclusion: 6 months Duration of patient's participation: one day

DETAILED DESCRIPTION:
According to the data of the French Health Insurance, near 40% of French people aged 65 years and over and suffering from Alzheimer disease and associated disorders (ADAD) are exposed to antidepressants (AD) versus 13% of those without ADAD. This confirms the international data on the prevalence of antidepressant prescription in people with ADAD ranging from 26% to 56.4% but always superior to those of the population with the same age.

If depression and anxiety disorders are comorbidities frequently associated with dementia, such level of AD exposure suggests an overuse of AD in this population. This overuse has been described in people living in nursing home (among those, a majority suffers from ADAD) and would reach 62%. To assess this overuse in demented people whatever their place of living is necessary to further implement risk minimization actions.

Hypothesis : Overuse of AD is frequent in patients with ADAD. It is possible to assess overuse associated with off label prescriptions (no validated indication and excess in the prescription duration) through a transversal study.

Main objective : To assess the prevalence of AD overuse associated with off label prescriptions (no validated indication and excess in the prescription duration) in patients aged 70 years and over with ADAD.

Secondary objectives :

1. To assess the prevalence of AD prescribed for a non validated indication
2. To assess the prevalence of AD prescribed with an excess in prescription duration
3. To assess the prevalence of psychotropic coprescription and notably the prevalence of the neurologic iatrogenic alerts as defined by the French National Authority for Health:

   * Any prescription of a long half-life benzodiazepine;
   * Of neuroleptics in Alzheimer patients; or
   * Of 3 or more psychotropic drugs)
4. To assess factors associated to AD overuse

Measurements : AD overuse with off label prescriptions, ie no validated indication or excess in prescription duration :

* Drug will be defined as AD if they are included in the list of AD designed by a national French Task Force including experts from over 30 associations and scientific societies (N06AA02 Imipramine, N06AA04 Clomipramine, N06AA06 Trimipramine, N06AA09 Amitriptyline, N06AA10 Nortriptyline, N06AA17 Amoxapine, N06AA21 Maprotiline, N06AB03 Fluoxetine, N06AB04 Citalopram, N06AB05 Paroxetine, N06AB06 Sertraline, N06AB08 Fluvoxamine, N06AB10 Escitalopram, N06AF03 Phenelzine, N06AF04 Tranylcypromine, N06AF05 Iproniazide, N06AG02 Moclobemide, N06AX03 Mianserine, N06AX11 Mirtazapine, N06AX14 Tianeptine, N06AX16 Venlafaxine, N06AX17 Milnacipran, N06AX21 Duloxetine, N06AX22 Agomelatine)
* Indication for AD will be the one declared by the prescriber of AD. This data will be collected through direct contact with prescriber or medical report or record or interview of patient's caregiver.
* Off label prescription will be defined by prescription for indication not listed in the Summary of Product Characteristics (SPC).
* Prescription duration will be considered as exceeded if superior to that recommended in market authorization:
* Duration>14 months in major depressive disorder and in patient with remission
* Exceeded duration according to the geriatrician in charge according to the multidisciplinary evaluation performed during the geriatric day hospital . If the geriatrician could not conclude, an expert committee (including a psycho-geriatrician and a geriatrician expert in drug) will adjudicate to the overuse or not of the AD.

Method : A transversal monocentric study in the geriatric day Bretonneau unit will be performed. Study will be proposed to all eligible patients (with non-opposition of the patient or of his legal representative to the collection of his personal data). Included people will have no supplementary clinical or complementary investigations.

Data collected routinely in geriatric day hospital include :

Data collected by nurse: socio-demographic data/ functional abilities (ADL IADL)/ professional caregiver at home/ weight,pulse, blood pressure, orthostatic hypotension/ Zarit scale/ NeuroPsychiatric Inventory Data collected by geriatrician : medical history, medication conciliation, clinical exam, screening for depression (miniGDS or Cornell scale according to theMiniMental Status MMS score > or <18), MMSif latest score>one year, Frontal assessment battery at bedside (FAB) Psychologic or psychiatric assessment as neuropsychometric assessment are performed according to the indication for the cause of the assessment in the geriatric day hospital .

The geriatrician in charge will have to systematically collect the indication and the history of the AD treatment.

At the end of the evaluation performed in the geriatric day unit, the geriatrician will have to conclude to the AD overuse or not associated with off label prescription. Doubtful case will be examined by a validation committee ( psychogeriatrician and geriatrician expert in drug).

Inclusion criteria : age ≥70 years / dementia according to DSMIV criteria, whatever its level/ Antidepressant prescription Non inclusion criteria: opposition of the patient or of his legal representative to the collection of his personal data/ Mild Cognitive Impairment Sample size Considering that 40% of people suffering from ADAD are prescribed antidepressant (data from French Health Insurance), the number of eligible patients consulting in the geriatric day swill be 65 in 6 months. If 10% of them are opposed to the collection of their personal data and if the overuse of AD is near 50% , precision of the result will be 12.8% (95%CI bilateral).

Duration of inclusion : 6 months. Duration of patient's participation : one day.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥70 years,
* Dementia according to DSMIV criteria, whatever its level,
* Antidepressant prescription.

Exclusion Criteria:

* Refusal of the patient or of his legal representative to the collection of his personal data,
* Mild Cognitive Impairment.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Seniors (age 70 or older) with dementia on antidepressants.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
AD overuse with off label prescriptions, ie no validated indication or excess in prescription duration. | At inclusion
  Indication for AD will be the one declared by the prescriber of AD. Off label prescription will be defined by prescription for indication not listed in the Summary of Product Characteristics (SPC).
  Prescription duration will be considered as exceeded if superior to that recommended in market authorization :
  Duration>14 months in major depressive disorder and in patient with remission Exceeded duration according to the geriatrician in charge according to the multidisciplinary evaluation performed during the geriatric day hospital . If the geriatrician could not conclude, an expert committee (including a psycho-geriatrician and a geriatrician expert in drug) will adjudicate to the overuse or not of the AD.

SECONDARY OUTCOMES:
Prevalence of psychotropic coprescription | At inclusion
  Prevalence of coprescription with antipsychotic, anxiolytic annd hypnotic
Prevalence of the neurologic iatrogenic alerts as defined by the French National Authority for Health | At inclusion
  Prevalence of coprescription of a long half-life benzodiazepine ; of neuroleptics and of 3 or more psychotropic drugs
Type and severity of dementia (Mini Mental Status, Frontal Assessment Battery, stage of dementia, etiological diagnosis) | At inclusion
  Type and severity of dementia (MMS "Mini Mental Status", FAB "Frontal Assessment Battery", stage of dementia : early stage ; early to middle ; middle ; middle to late ; late stage, etiological diagnosis : Alzheimer's dementia, vascular dementia, both Alzheimer's disease and vascular dementia, another form of dementia (please precise), unknown etiology)
Comorbidities | At inclusion
Coprescription, type and number of prescriber(s) | At inclusion
Type and number of help at home (professional and non professional caregivers) | At inclusion
Non-drug therapy in conjunction with anti-depressant medication : yes or no (if yes, please name the therapy) | At inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Dominique BONNET-ZAMPONI, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Bretonneau, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided